CLINICAL TRIAL: NCT02788019
Title: Adductor Canal Mid-thigh and Adductor Canal Distal Thigh: Is Cutaneous Sensory Blockade Similar Among Block Techniques?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to complete the sample size needed for 80% power due to changes in surgical approach to adductor block usage.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Machi, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 092015-065
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
Keywords: Adductor canal block, nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mid-Thigh Adductor Block (Experimental): Subject will receive a mid-thigh adductor block method using ropivacaine (0.5%, 15 mL).
  Interventions: Drug: Ropivacaine
- Distal-Thigh Adductor Block (Active Comparator): Subject will receive a distal-thigh adductor block method using ropivacaine (0.5%, 15 mL).
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine is routinely used to perform localized blockade prior to surgery to improve management of postoperative pain.

SUMMARY:
This is a randomized noninferiority interventional study to determine the equivalence of two adductor canal block (ACB) methods: mid-thigh and distal thigh in patients undergoing medial foot, medial ankle, or medial leg surgery. Sixty eight patients will be identified during their orthopedic presurgical clinic visit, anesthesia preoperative clinic visit or Day Surgery Unit (Zale Lipshy Hospital, Clements University Hospital, and University of Texas Southwestern Outpatient Surgery Center) for eligibility. Eligible individuals may be introduced to the study in the orthopedic presurgical clinic or the anesthesia preoperative clinic by staff. After consent patients will be randomized (break-seal method) to receive either a mid-thigh or distal thigh block using ropivacaine prior to foot, ankle, or leg surgery. The following measurements will be obtained to determine the change in sensory distribution: pinprick test with Neuropen, maximum voluntary isometric contraction before and after block, postoperative pain scores (24 hrs and at discharge) and postoperative opiate consumption.

DETAILED DESCRIPTION:
Potential subjects will be identified at the orthopedic presurgical clinic, the anesthesia preoperative clinic or the Day Surgery Unit. The electronic medical record (Epic) will also be used for prescreening potential subjects. Recruitment and consenting at will occur at anesthesia preoperative clinics, Day Surgery Unit. A computer generated randomization list will be used for randomization list. The research intervention of this study will take place within the standard clinical context. The patient will receive an ACB regardless of their participation in this research in accordance with their anesthetic plan and their desires The experiment will be conducted as follows: A 20-point grid will be drawn on the subject's leg that will receive medial foot, ankle or leg surgery. Two baseline measurements will be taken prior to administration of the adductor block: distribution of sensation using pinprick (Neuropen) method, and muscle contraction strength using a dynamometer. The number of grid cells with sensation will be counted and recorded. The randomized block will be administered allowing 20 minutes for anesthetic to take full effect. Post-block measurements include pinprick in each of the grid cells, where patient will indicate whether sensation is felt or not. The cells where sensation is perceived will be circled and number of cells will be recorded. After sensation is recorded, maximum voluntary isometric contraction (MVIC) will again be measured with the dynamometer to record the maximal contraction strength. Within 24 hours of surgery, the subject will be asked to rate their pain on a scale of 0-10, and will be recorded again after discharge, in conjunction with opiates required to reduce pain. A more detailed explanation of experimental steps can be read below.

20-Point Grid: The 20-point grid will be marked starting with anatomical landmarks at the knee joint: the medial inter-knee joint where the tibia meets the femur, the mid medial patella, the mid lateral patella, and along the same line at the semitendinosus tendon at 5 cm posterior from that point. Then 5 cm intervals will be plotted progressing cephalad to a total of 15 cm.

Neuropen test:

Prior to administration of randomized blockade technique a pinprick test will be administered using a Neuropen on a scale of 0-1, with 1-normal sharp sensation and 0=dull change of sensation. Mechanical stimulation with pinprick testing is routinely used to test nociception in the bedside neurologic examination. Sharpness can be considered a surrogate for nociception because whereas sharpness is not necessarily painful, mechanical thresholds for sharpness closely parallel those for pain. The subject will be asked to determine whether the stimulus feels sharp. The number of grid-points with a change in sensation from baseline will be recorded at baseline and 20 minutes after the block.

MVIC:

Additionally, MVIC will be measured by a handheld dynamometer (Lafayette Instrument Company, Lafayette Indiana) to determine muscle strength at baseline and after the adductor block. The patient will be in a seated position with the thigh parallel to the floor and the knee at a 90-degree angle with the feet off the floor. The dynamometer is applied to the leg 5 cm above the transmalleolar axis and perpendicular to the tibial crest. The patient is instructed to extend the leg at the knee with sustained maximal force for 5 seconds. This will be repeated 3 times with 30 seconds rest between each movement, and the force will be recorded (Newtons).

Adductor Canal Blockade The adductor canal block will be performed using a linear HFL38xp or a linear HFL38x ultrasound probe (X-Porte or M-Turbo; SonoSite; Bothell, Washington). The site that is to receive the ACB will be sterilized with chlorhexidine gluconate 2% and 70% isopropyl alcohol prep. A skin weal of lidocaine 1% (2-5mL) will be delivered. A Tuohy needle (17 gauges) will be inserted through the skin wheal under ultrasound guidance towards the target nerve location. Ropivacaine 0.5% 15ml will be injected for either adductor canal locations.27 Pain Scores and Opiate Consumption A follow-up visit will be performed in person for inpatients or via phone for outpatients within 24 hours from discharge to assess for pain control, and monitoring side effects. It will take 10 minutes. Adverse events will be monitored during the 24-hour period of the study.

Potential Risks Potential risks include loss of confidentiality or mild discomfort associated with the pinprick for sensory testing. Risks that are involved with administration of ropivacaine are primarily damage to surrounding tissues, including nerves, and may cause bleeding or infection from injection or an unknown allergy to ropivacaine that develops during the administration of the drug. There are no additional physical or psychological risks that may result from participation in this research protocol since patients will have determined that they desire perineural blockade before study inclusion is even proposed.

Subject Safety and Data Monitoring Any serious adverse reaction, including allergy and local anesthetic systemic toxicity, will result in immediate discontinuation of study related procedures and treatment as necessary. Serious adverse events will be reported to the Institutional Review Board. The data already obtained from a participant who has had a serious adverse event will be analyzed according to intention-to-treat principle.

If non-inferiority between the two neurosensory blockade techniques is significantly detected at 50% enrollment (or enrollment of 34 patients), the study will be stopped. The study will also be stopped in the event that there is overwhelming statistical evidence at interim analysis that the two blocks are different, or in the very small chance that there are multiple adverse events in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Individuals undergoing surgery of the medial foot, medial ankle, or medial leg for which the anesthetic plan includes an adductor canal nerve block

Exclusion Criteria:

1. Any known deficit of the ipsilateral lumbar nerve roots, ipsilateral lumbar plexus, ipsilateral femoral nerve, obturator nerve or saphenous nerve including diabetic peripheral neuropathy
2. Any local disorder of the skin or otherwise where blockade is to be performed
3. Body mass index >50
4. American Society of Anesthesiologists (ASA) classification greater than 3
5. Allergy to amide local anesthetic medications
6. Pregnancy
7. Incarceration
8. Inability to understand study procedures including inability to understand the English language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Machi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Zale Lipshy University Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Tubbs RS, Loukas M, Shoja MM, Apaydin N, Oakes WJ, Salter EG. Anatomy and potential clinical significance of the vastoadductor membrane. Surg Radiol Anat. 2007 Oct;29(7):569-73. doi: 10.1007/s00276-007-0230-4. Epub 2007 Jul 7. PMID 17618402
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Machi AT, Sztain JF, Kormylo NJ, Madison SJ, Abramson WB, Monahan AM, Khatibi B, Ball ST, Gonzales FB, Sessler DI, Mascha EJ, You J, Nakanote KA, Ilfeld BM. Discharge Readiness after Tricompartment Knee Arthroplasty: Adductor Canal versus Femoral Continuous Nerve Blocks-A Dual-center, Randomized Trial. Anesthesiology. 2015 Aug;123(2):444-56. doi: 10.1097/ALN.0000000000000741. PMID 26079800
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Defining adductor canal block. Reg Anesth Pain Med. 2014 May-Jun;39(3):253-4. doi: 10.1097/AAP.0000000000000052. No abstract available. PMID 24747312
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Redefining the adductor canal block. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):442-3. doi: 10.1097/AAP.0000000000000119. No abstract available. PMID 25140514
- [Background] Jaeger P, Lund J, Jenstrup MT, Brondum V, Dahl JB. Reply to Dr Bendtsen. Reg Anesth Pain Med. 2014 May-Jun;39(3):254-5. doi: 10.1097/AAP.0000000000000069. No abstract available. PMID 24747313
- [Background] Cowlishaw P, Kotze P. Adductor canal block--or subsartorial canal block? Reg Anesth Pain Med. 2015 Mar-Apr;40(2):175-6. doi: 10.1097/AAP.0000000000000205. No abstract available. PMID 25688724
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. Basic Topography of the Saphenous Nerve in the Femoral Triangle and the Adductor Canal. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):391-2. doi: 10.1097/AAP.0000000000000261. No abstract available. PMID 26079358
- [Background] Benzon HT, Sharma S, Calimaran A. Comparison of the different approaches to saphenous nerve block. Anesthesiology. 2005 Mar;102(3):633-8. doi: 10.1097/00000542-200503000-00023. PMID 15731603
- [Background] Lopez AM, Sala-Blanch X, Magaldi M, Poggio D, Asuncion J, Franco CD. Ultrasound-guided ankle block for forefoot surgery: the contribution of the saphenous nerve. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):554-7. doi: 10.1097/AAP.0b013e3182611483. PMID 22854395
- [Background] Backonja MM, Walk D, Edwards RR, Sehgal N, Moeller-Bertram T, Wasan A, Irving G, Argoff C, Wallace M. Quantitative sensory testing in measurement of neuropathic pain phenomena and other sensory abnormalities. Clin J Pain. 2009 Sep;25(7):641-7. doi: 10.1097/AJP.0b013e3181a68c7e. PMID 19692807
- [Background] Kocarev M, Watkins E, McLure H, Columb M, Lyons G. Sensory testing of spinal anaesthesia for caesarean section: differential block and variability. Int J Obstet Anesth. 2010 Jul;19(3):261-5. doi: 10.1016/j.ijoa.2010.02.002. Epub 2010 Jun 2. PMID 20627691
- [Background] Maffiuletti NA. Assessment of hip and knee muscle function in orthopaedic practice and research. J Bone Joint Surg Am. 2010 Jan;92(1):220-9. doi: 10.2106/JBJS.I.00305. PMID 20048117
- [Background] Lu YM, Lin JH, Hsiao SF, Liu MF, Chen SM, Lue YJ. The relative and absolute reliability of leg muscle strength testing by a handheld dynamometer. J Strength Cond Res. 2011 Apr;25(4):1065-71. doi: 10.1519/JSC.0b013e3181d650a6. PMID 20838248
- [Background] Reinking MF, Bockrath-Pugliese K, Worrell T, Kegerreis RL, Miller-Sayers K, Farr J. Assessment of quadriceps muscle performance by hand-held, isometric, and isokinetic dynamometry in patients with knee dysfunction. J Orthop Sports Phys Ther. 1996 Sep;24(3):154-9. doi: 10.2519/jospt.1996.24.3.154. PMID 8866274
- [Background] Walk D, Sehgal N, Moeller-Bertram T, Edwards RR, Wasan A, Wallace M, Irving G, Argoff C, Backonja MM. Quantitative sensory testing and mapping: a review of nonautomated quantitative methods for examination of the patient with neuropathic pain. Clin J Pain. 2009 Sep;25(7):632-40. doi: 10.1097/AJP.0b013e3181a68c64. PMID 19692806
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study patients were followed after block procedure for 24 hrs. Adverse events were also monitored within this period.
Period: Overall Study
Arm/Group | Mid-Thigh Adductor Block | Distal-Thigh Adductor Block
Started | 27 | 25
Completed | 23 | 20
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: The study was terminated for failure of enrollment prior to reaching 34 participants in each group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mid-Thigh Adductor Block | Distal-Thigh Adductor Block | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.62 (15.02) | 57.84 (12.37) | 57.21 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 25 | 52
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28.5 [25.8 to 35.0] | 30.9 [24.4 to 34.7] | 29.8 [24.95 to 34.85]

OUTCOME MEASURES:

1. Primary Outcome: Number of Grid Points With Change of Sensation to Pinprick After Blockade
Description: The distribution of cutaneous sensation affected by the different techniques of adductor canal blockade is assessed using a monofilament Neuropen to prick points on a 20 point grid applied to the skin in a standard fashion according to this method: A grid will be marked starting with anatomical landmarks at the knee joint: the medial inter-knee-joint point where the tibia meets the femur, the mid medial patella, the mid lateral patella, and along the same line at the semitendinosus tendon and 5cm posterior from that point. Then 5cm intervals will be plotted progressing cephalad to a total of 15 centimeters. This will yield 20 grid points (5x4 points). Once the grid is made, testing proceeds with a Neuropen on a scale of 0-1, with 1 = normal sharp sensation, 0 = change of sensation. The Neuropen is used for the standardization of force.
Time Frame: 20 minutes
Population: Only patients who were enrolled and had data for both pre and post blockade were considered for this analysis.
Measure: Mean (Standard Deviation); unit: points of cutaneous sensation
Arm/Group | Mid-Thigh Adductor Block | Distal-Thigh Adductor Block
Number analyzed (Participants) | 27 | 25
points of cutaneous sensation | 19.81 (0.55) | 20 (0)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from the time point of receiving an adductor block up to 24 hrs post block.
Description: We used an electronic version of the National Center for Complementary and Integrative Health (United States National Institutes of Health) adverse collection form.
Arm/Group | Mid-Thigh Adductor Block | Distal-Thigh Adductor Block
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 1/27 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid-Thigh Adductor Block (N=27) | Distal-Thigh Adductor Block (N=25)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient developed herpes zoster lesions on flank of the side he received his block in.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT02788019/Prot_SAP_000.pdf